CLINICAL TRIAL: NCT00908453
Title: The Study of NPC-06 - Investigation of Safety, Efficacy and Pharmacokinetics of Fosphenytoin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Nobelpharma Co., Ltd., CNS group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-06-2
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Epilepsy
Keywords: NPC-06; fosphenytoin; phenytoin; pharmacokinetics; safety
MeSH Terms: conditions — Epilepsy | interventions — fosphenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 15mg/kg of loading dose (Experimental)
  Interventions: Drug: fosphenytoin
- 18mg/kg of loading dose (Experimental)
  Interventions: Drug: fosphenytoin
- 22.5mg/kg of loading dose (Experimental)
  Interventions: Drug: fosphenytoin

INTERVENTIONS:
Drug: fosphenytoin — 15mg/kg, 18mg/kg or 22.5mg/kg of loading doses of fosphenytoin

SUMMARY:
The study is to evaluate safety, efficacy and pharmacokinetics of intravenously administered fosphenytoin in patients with neurosurgery, head trauma, epilepsy or status epilepticus who are requiring a loading dose of phenytoin.

ELIGIBILITY:
Inclusion Criteria:

* male or female, hospitalized patients 2 years of age or older
* Adult patients or guardian for pediatric patients to provide written informed consent

Exclusion Criteria:

* patient with a history of hypersensitivity to hydantoins
* patient with hypotension, sinus bradycardia, sino-atrial block, second or third degree A-V block, or Adams-Stokes syndrome
* pregnant or nursing female patients

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 8 to 12 days

SECONDARY OUTCOMES:
frequency and nature of seizures | 8 to 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Nakagawa, M.D., Study Director — National Center of Neurology and Psychiatry
Locations (1):
- National Center of Neurology and Psychiatry, Kodaira, Tokyo, Japan